CLINICAL TRIAL: NCT03360279
Title: A Randomized Trial Comparing Drug-coated Balloon and Regular Balloon for Dialysis Access Stent Graft Restenosis
Brief Title: DCB for Dialysis Access Stent Graft Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, IRB of NTUH Hsin-Chu Branch, Mu-Yang Hsieh MD, National Taiwan University Hospital Hsin-Chu Branch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105-015-F
Record Dates: First submitted 2017-11-12; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Hemodialysis Access Failure (Disorder); Stent-Graft Restenosis; Arteriovenous Graft; Drug-coated Balloon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The IVUS interpreter and follow-up evaluators are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular balloon (Active Comparator): Use the regular balloon to perform standard balloon angioplasty.
  Interventions: Device: Regular balloon
- DCB (paclitaxel-coated balloon) (Active Comparator): Use DCB (paclitaxel-coated balloon) to perform additional balloon angioplasty.
  Interventions: Device: DCB (paclitaxel-coated balloon)

INTERVENTIONS:
Device: Regular balloon — Randomization: to use regular balloon to treat stent graft restenosis
  Arms: Regular balloon
Device: DCB (paclitaxel-coated balloon) — Randomization: to use DCB (paclitaxel-coated balloon, Ranger, Boston-Scientific) to treat stent graft restenosis. The paclitaxel dose is 2 ug/mm2 delivered with the Ranger drug-coated balloon.
  Arms: DCB (paclitaxel-coated balloon)

SUMMARY:
Recurrent stenosis in hemodialysis access graft (AVG) is difficult to treat. For recurrent stenosis in the anastomotic junction can be treated by stent graft to improve long-term patency. However, there is no data regarding treatment of stent graft restenosis in AVG. This randomized trial is designed to compare the efficacy and safety of drug-coated balloon (DCB) versus regular balloon in AVG stent graft restenosis.

DETAILED DESCRIPTION:
Prosthetic arteriovenous hemodialysis access graft (AVG) has high incidences of venous anastomotic stenosis and access failure. A stent graft can be used in AVG with recurrent venous anastomotic stenosis to improve long-term patency rate. However, after stent graft implementation, the effective treatment for restenosis in a stent graft is still unknown. This randomized trial is designed to evaluate the efficacy and safety of drug-coated balloon versus regular balloon for in-stent restenosis in stent graft. The investigators plan to enroll 40 patients who presented with prosthetic AVG in-stent restenosis, and then to evaluate the restenosis lesions by intravascular ultrasound. Patients will be randomized into two groups of treatment: drug-coated balloon angioplasty or regular balloon angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 to 90 years on regular hemodialysis at least 3 months
* Had stent graft implemented at dialysis vascular access
* Angiographic evidence of stenosis within the stent graft or less than 2 cm from the stent graft edge
* Clinical evidence of a hemodynamically significant stenosis or thrombosis
* Patient is able to provide written informed consent

Exclusion Criteria:

* Elbow fracture or any disease involve the elbow joint that prohibits the flexion maneuver.
* Target lesion cannot be crossed by the guide wire.
* Known hypersensitivity to heparin or contrast medium.
* Bleeding diathesis.
* Patients participating in another clinical trial with interfering with this trial in the past three months.
* Untreatable bleeding diathesis.
* Other diseases, such as cancer, liver disease, or cardiac insufficiency, which may lead to protocol violations or markedly shorten a patient's life expectancy (less than 3 months).
* Patients unable or unwilling to participate this trial.
* Pregnancy, lactating woman, non-adult, criminals in sentence, psychiatric patients, research staffs or colleagues are prohibited.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss | 0, 1, and 3 months
  The late luminal loss found by IVUS on follow-up in comparison to index procedure.

SECONDARY OUTCOMES:
minimal luminal area and diameter | 0, 1, and 3 months
  Done by IVUS on follow-up in comparison to index procedure.
restenosis rate | 0, 1, and 3 months
  Compare with follow-up angiography.
repeated intervention | 0, 1, and 3 months
  defined by repeated endovascular balloon angioplasty or endovascular thrombectomy or surgical open thrombectomy.
abandon of AV graft, death | 0, 1, and 3 months
  stopped to use the target AVG or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Yang Hsieh, MD, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Hsinchu City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsieh MY, Lin PS, Liao MT, Lin L, Chen TY, Boon JC, Yang TF, Wu CC. A Randomised Trial Comparing Drug Coated Balloons and Conventional Balloons for the Treatment of Stent Graft Stenosis in Dialysis Vascular Access. Eur J Vasc Endovasc Surg. 2023 Aug;66(2):253-260. doi: 10.1016/j.ejvs.2023.05.028. Epub 2023 May 18. PMID 37209996

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03360279/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03360279/ICF_001.pdf